CLINICAL TRIAL: NCT00439335
Title: A Phase I/II Randomized, Double-Blinded Placebo-Controlled Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of Immunization With Inactivated Subvirion Influenza A/H5N1 Vaccine Administered by the Intradermal or the Intramuscular Route Among Healthy Adults
Brief Title: Higher Dose Intradermal H5 Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-0089
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2009-05-08 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2009-08

CONDITIONS: Influenza
Keywords: Influenza, vaccine, A/H5N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- H5 HA IM (Experimental): Vaccine group H5 HA IM: the subject will receive 0.1 mL of H5 HA by the IM route in one arm and 0.1 mL of saline placebo by the ID route in the other arm.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1; Drug: Placebo (ID)
- H5 HA ID (Experimental): Vaccine group H5 HA ID: the subject will receive 0.1 mL of H5 HA by the ID route in one arm and 0.1 mL of saline placebo by the IM route in the other arm.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1; Drug: Placebo (IM)

INTERVENTIONS:
Biological: Inactivated Influenza A Vaccine A/H5N1 — Inactivated influenza A/H5N1 vaccine formulated to a concentration of HA greater than or equal to 300 mcg/mL administered via intramuscular (IM) injection. Vaccine will be administered to each subject at Days 0 and 28.
  Arms: H5 HA IM
Biological: Inactivated Influenza A Vaccine A/H5N1 — Inactivated influenza A/H5N1 vaccine formulated to a concentration of HA greater than or equal to 300 mcg/mL administered via intradermal (ID) injection. Vaccine will be administered to each subject at Days 0 and 28.
  Arms: H5 HA ID
Drug: Placebo (IM) — The placebo will be 0.1 mL of saline administered by the IM route.
  Arms: H5 HA ID
Drug: Placebo (ID) — The placebo will be 0.1 mL of saline administered by the ID route.
  Arms: H5 HA IM

SUMMARY:
This study will compare the influenza A/H5N1 virus vaccine given by injection in the muscle versus injection in the skin in healthy adults. The study will look at the safety of the injections, how the body reacts, and what the body's immune response does when the vaccine is given in the muscle versus in the skin. The study will look at 226 healthy volunteers, ages 18-49 years old. Study procedures will include getting 2 doses of vaccine 28 days apart, physical exams, follow-up clinic visits to check the places on the body where each vaccine was given, and blood sample collections. Volunteers will complete a memory aid by writing down temperatures and health changes for 7 days after each vaccination. Volunteers will be involved in the study for up to 241 days.

DETAILED DESCRIPTION:
Influenza A viruses have the potential to cause worldwide epidemics and/or pandemics resulting in significant morbidity and mortality. Two-hundred twenty-six healthy male and female subjects aged 18 to 49 years, inclusive, in the United States (US) will be enrolled into this single-center, randomized, double-blinded, placebo-controlled trial of intradermal (ID) and intramuscular (IM) injection with subvirion (SV) inactivated influenza A/H5N1 vaccine. The study will have two vaccine groups. Vaccine group 1: the subject will receive 0.1 mL of H5 Hemagglutination (HA) by the ID route in one arm and 0.1 mL of saline placebo by the IM route in the other arm. Vaccine group 2: the subject will receive 0.1 mL of H5 HA by the IM route in one arm and 0.1 mL of saline placebo by the ID route in the other arm. All eligible subjects will be enrolled and randomized 1:1 (113 subjects per vaccine group) to either vaccine group 1 or vaccine group 2. All subjects will receive two doses of approximately 30micrograms of H5 HA by their assigned route, either IM or ID, separated by approximately 28 days. At each vaccination visit, all subjects will also receive a saline placebo in the opposite arm by the different route as their vaccine route (i.e. if vaccine is administered by the ID route in one arm, then a saline placebo will be administered by the IM route in the opposite arm). The second vaccine dose will be administered by the same route as per vaccine group assigned at original randomization. Subjects will be observed in the clinic for approximately 15 minutes after each vaccination. Subjects will return on Day 2 for arm check and assessment of adverse events. All subjects will maintain a memory aid recording oral temperature, and systemic and local adverse events for 7 days after each vaccination. They will return to clinic on Day 8 for adverse event (AE) assessment, concomitant medication assessment, a targeted physical exam (if indicated), and review of memory aid. AE data will be captured Day 0 through Day 56. Serious AE data will be captured from Day 0 through the end of each subject's participation in the study (approximately 7 months). The subjects, staff assessing subjects, and lab personnel will be blinded. Serum for immunogenicity evaluations will be obtained prior to the first vaccination, at Day 0; prior to the second vaccination, at Day 28; on Day 56 and approximately Day 208 (7months after dose 1). The primary objectives are to compare the immunogenicity of a similar dosage level of a subvirion inactivated influenza A/H5N1 vaccine given by ID or IM injection one month after receipt of the second dose of vaccine and to compare the safety and reactogenicity of ID and IM immunization at a similar dosage level of a subvirion inactivated influenza A/H5N1 vaccine among healthy young adults. The secondary objective is to evaluate serum antibody responses approximately 1 and 7 months after the first vaccination. This study is linked to Division of Microbiology and Infectious Diseases protocol 07-0022.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female between the ages of 18 and 49 years, inclusive.
* Women of childbearing potential (not surgically sterile or post menopausal for greater than or equal to 1 year) must agree to practice adequate contraception (i.e., barrier method, abstinence, intrauterine devices, or licensed hormonal methods) for the entire study period.
* Is in good health, as determined by vital signs (heart rate less than 100 beats per minute; blood pressure: systolic less than or equal to 140 mm Hg and greater than or equal to 90 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature less than 100.0 degrees Fahrenheit), medical history to ensure stable medical condition (see definition below) and a targeted physical examination based on medical history.

Stable medical condition - no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.

* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine.
* Has a positive urine or serum pregnancy test prior to vaccination (if female of childbearing potential), is breastfeeding, or has the intention to become pregnant during the study period.
* Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Long term use of oral or parenteral steroids, high-dose inhaled steroids (greater than 800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Has a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Has been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Is receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has a moderate to severe acute illness and/or an oral temperature greater than 100.4 degrees Fahrenheit, within 1 week of vaccination.
* Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the 5 years prior to enrollment.
* Presence of any active skin disease on upper arms that could impact study product delivery or site assessment.
* Has a history of Guillain Barre syndrome.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expects to receive an experimental agent during the 7-month study period.
* Participated in an Influenza A/H5 vaccine study in the past in a group receiving vaccine (but does not exclude documented placebo recipients).
* Is enrolled or planning to enroll in another interventional trial at any time between receipt of the first dose of vaccine and the end of the study (approximately 7 months after receipt of the first dose).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Patel SM, Atmar RL, El Sahly HM, Guo K, Hill H, Keitel WA. Direct comparison of an inactivated subvirion influenza A virus subtype H5N1 vaccine administered by the intradermal and intramuscular routes. J Infect Dis. 2012 Oct 1;206(7):1069-77. doi: 10.1093/infdis/jis402. Epub 2012 Aug 13. PMID 22891287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy ambulatory adults were recruited from the surrounding community of the research clinic from March 14, 2007 to June 20, 2007.
Period: Overall Study
Arm/Group | H5 HA ID | H5 HA IM
Started | 113 | 114
Completed | 111 | 114
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H5 HA ID | H5 HA IM | Total
Number analyzed (Participants) | 113 | 114 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 114 | 227
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (7.4) | 30.5 (8.0) | 30.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 60 | 134
  Male | 39 | 54 | 93
Region of Enrollment [Number; unit: participants]
  United States | 113 | 114 | 227

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a 4-fold or Greater Increase in HAI Antibody Titers After Dose 2
Description: Number of participants in each vaccine group achieving a 4-fold or greater increase in serum hemagglutination inhibition (HAI) antibody titers against influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine
Time Frame: Approximately Day 56.
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 113
Participants | 47 | 40

2. Primary Outcome: Number of Participants Spontaneously Reporting Any Serious Adverse Event.
Description: Any untoward medical occurrence that resulted in death, persistent/significant disability/incapacity, required in-patient hospitalization or prolongation thereof, was life threatening or a congenital anomaly/birth defect in offspring of a study subject; or may have jeopardized the participant or required intervention to prevent one of the outcomes.
Time Frame: Through Day 208.
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Participants | 2 | 2

3. Secondary Outcome: HAI Geometric Mean Titer (GMT) After Dose 2
Description: HAI geometric mean titer (GMT) against influenza A/H5N1 virus in each vaccine group 28 days after receipt of the second dose of vaccine.
Time Frame: Approximately Day 56.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody Titer
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 113
Antibody Titer | 25.2 [18.3 to 34.5] | 18.1 [13.6 to 24.1]

4. Secondary Outcome: Number of Participants Achieving a HAI Titer of Greater Than or Equal to 40 After Dose 2
Description: Number of participants achieving a serum HAI titer of greater than or equal to 40 against influenza A/H5N1 virus in each vaccine group 28 days after receipt of the second dose of vaccine
Time Frame: Approximately Day 56
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 113
Participants | 48 | 40

5. Secondary Outcome: Number of Participants Achieving a 4-fold or Greater Increase in HAI Antibody Titers After Dose 1.
Description: Number of participants achieving a 4-fold or greater increase in HAI antibody titers against influenza A/H5N1 virus in each vaccine group one month after receipt of the first dose.
Time Frame: Approximately Day 28
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Participants | 25 | 29

6. Secondary Outcome: HAI GMT After Dose 1
Description: HAI GMT against influenza A/H5N1 virus one month after receipt of the first dose of vaccine.
Time Frame: Approximately Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody titer
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Antibody titer | 13.1 [9.9 to 17.3] | 11.9 [9.1 to 15.4]

7. Secondary Outcome: Number of Participants Achieving a Serum HAI Titer of Greater Than or Equal to 40 After Dose 1.
Description: Number of participants achieving a serum HAI titer of greater than or equal to 40 against influenza A/H5N1 virus in each vaccine group one month after receipt of the first dose of vaccine.
Time Frame: Approximately Day 28
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Participants | 26 | 29

8. Secondary Outcome: Number of Participants Achieving a 4-fold or Greater Increase in HAI Antibody Titers 7 Months After Dose 1.
Description: Number of participants achieving a 4-fold or greater increase in HAI antibody titers against influenza A/H5N1 virus in each vaccine group seven months after receipt of the first dose of vaccine.
Time Frame: Approximately Day 208
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 111 | 112
Participants | 17 | 16

9. Secondary Outcome: HAI GMT at 7 Months After Dose 1
Description: HAI GMT against influenza A/H5N1 virus in each vaccine group seven months after receipt of the first dose of vaccine.
Time Frame: Approximately Day 208
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody Titer
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 111 | 112
Antibody Titer | 10.0 [8.1 to 12.4] | 8.9 [7.3 to 10.9]

10. Secondary Outcome: Number of Participants Achieving a Serum HAI Titer of Greater Than or Equal to 40 at 7 Months After Dose 1.
Description: Number of participants achieving a serum HAI titer of greater than or equal to 40 against influenza A/H5N1 virus in each vaccine group 7 months after receipt of the first dose of vaccine.
Time Frame: Approximately Day 208
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 111 | 112
Participants | 20 | 16

11. Primary Outcome: Occurrence of Unsolicited Symptoms During a 28-day Surveillance Period Following Vaccinations at Days 0 and 28.
Description: The number of participants spontaneously reporting any symptom (defined as any Adverse Event considered associated with the product) within 28 days of vaccination. Participants are counted only once but may have experienced events on multiple occasions.
Time Frame: Through approximately Day 56
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 113
Participants | 39 | 26

12. Primary Outcome: Occurrence of Solicited Systemic Symptoms During a 7-day Surveillance Period (Systematically Collected) Following Vaccinations at Days 0 and 28.
Description: The number of participants reporting fever, feverishness, malaise, myalgia, headache and nausea. Participants are counted only once for each symptom but may have experienced symptoms on multiple occasions.
Time Frame: 7 days after each vaccination
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Participants
  Fever | 2 | 2
  Feverishness | 11 | 14
  Malaise | 40 | 39
  Myalgia | 19 | 23
  Headache | 53 | 45
  Nausea | 14 | 13

13. Primary Outcome: Occurrence of Solicited Local Symptoms During a 7-day Surveillance Period (Systematically Collected) Following Vaccinations at Days 0 and 28.
Description: The number of participants reporting pain, tenderness, itching, induration, erythema, and pigmentation. Participants are counted only once for each symptom but may have experienced symptoms on multiple occasions.
Time Frame: 7 days after each vaccination
Measure: Number; unit: Participants
Arm/Group | H5 HA ID | H5 HA IM
Number analyzed (Participants) | 113 | 114
Participants
  Pain | 23 | 61
  Tenderness | 93 | 91
  Itching | 95 | 8
  Induration | 113 | 34
  Erythema | 113 | 59
  Pigmentation | 70 | 2

ADVERSE EVENTS:
Time Frame: Subjects recorded solicited symptoms on a memory aid for 8 days (Day 0-7) following each dose. Unsolicited non-serious adverse events were collected for 28 days after each dose and serious adverse events were collected through Day 208.
Description: The solicited symptoms are reported separately after each vaccination. The occurrence of a solicited symptom on any day(s) at any severity within the 15 day period was considered one event.
Arm/Group | H5 HA ID | H5 HA IM
Serious Adverse Events (participants affected / at risk) | 2/113 | 2/114
Other Adverse Events (participants affected / at risk) | 113/113 | 114/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H5 HA ID (N=113) | H5 HA IM (N=114)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Insulin-requiring type II diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | H5 HA ID (N=113) | H5 HA IM (N=114)
Injection site bruising (General disorders) | 13 (14) | 13 (13)
Injection site desquamation (General disorders) | 9 (11) | 1 (1)
Reactogenicity event (General disorders) | 113 (541) | 9 (10)
Hypersensitivity (Immune system disorders) | 7 (9) | 2 (2)
Gastroenteritis (Infections and infestations) | 7 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 19 (19)
Headache (Nervous system disorders) | 9 (10) | 14 (17)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (6) | 6 (7)
Injection site erythema - post dose 1 (General disorders) | 113 (113) | 42 (42) — Solicited on the memory aid as "Erythema (redness)" and measured in millimeters.
Injection site erythema - post dose 2 (General disorders) | 113 (113) | 42/113 (42) — Solicited on the memory aid as "Erythema (redness)" and measured in millimeters.
Injection site induration (size) - post dose 1 (General disorders) | 113 (113) | 20 (20) — Solicited on the memory aid as "Induration (swelling)" and measured in millimeters.
Injection site induration (size) - post dose 2 (General disorders) | 113 (113) | 23/113 (23) — Solicited on the memory aid as "Induration (swelling)" and measured in millimeters.
Injection site induration (functional grading) - post dose 1 (General disorders) | 113 (113) | 20 (20) — Solicited on the memory aid as "Induration (swelling)" with grading based on impact on daily activities.
Injection site induration (functional grading) - post dose 2 (General disorders) | 113 (113) | 24/113 (24) — Solicited on the memory aid as "Induration (swelling)" with grading based on impact on daily activities.
Injection site discolouration - post dose 1 (General disorders) | 37 (37) | 2 (2) — Solicited on the memory aid as "Pigmentation (discoloration)" and measured in millimeters.
Injection site discolouration - post dose 2 (General disorders) | 63 (63) | 0/113 (0) — Solicited on the memory aid as "Pigmentation (discoloration)" and measured in millimeters.
Injection site pruritus - post dose 1 (General disorders) | 80 (80) | 3 (3) — Solicited on the memory aid as "Itchiness at vaccination site"
Injection site pruritus - post dose 2 (General disorders) | 83 (83) | 7/113 (7) — Solicited on the memory aid as "Itchiness at vaccination site"
Injection site pain - post dose 1 (General disorders) | 18 (18) | 37 (37) — Solicited on the memory aid as "Pain at injection site at rest"
Injection site pain - post dose 2 (General disorders) | 10 (10) | 39/113 (39) — Solicited on the memory aid as "Pain at injection site at rest"
Tenderness - post dose 1 (General disorders) | 83 (83) | 79 (79) — Solicited on the memory aid as "Tenderness at injection site with movement/touch"
Tenderness - post dose 2 (General disorders) | 76 (76) | 67/113 (67) — Solicited on the memory aid as "Tenderness at injection site with movement/touch"
Feeling hot - post dose 1 (General disorders) | 8 (8) | 7 (7) — Solicited on the memory aid as "Feverishness"
Feeling hot - post dose 2 (General disorders) | 6 (6) | 8/113 (8) — Solicited on the memory aid as "Feverishness"
Headache - post dose 1 (Nervous system disorders) | 41 (41) | 36 (36) — Solicited on the memory aid as "Headache"
Headache - post dose 2 (Nervous system disorders) | 28 (28) | 20 (20) — Solicited on the memory aid as "Headache"
Malaise - post dose 1 (General disorders) | 32 (32) | 33 (33) — Solicited on the memory aid as "Malaise(decreased energy)"
Malaise - post dose 2 (General disorders) | 19 (19) | 19/113 (19) — Solicited on the memory aid as "Malaise(decreased energy)"
Myalgia - post dose 1 (Musculoskeletal and connective tissue disorders) | 15 (15) | 21 (21) — Solicited on the memory aid as "Myalgia - (body aches not at injection site)"
Myalgia - post dose 2 (Musculoskeletal and connective tissue disorders) | 8 (8) | 7/113 (7) — Solicited on the memory aid as "Myalgia - (body aches not at injection site)"
Nausea - post dose 1 (Gastrointestinal disorders) | 9 (9) | 9 (9) — Solicited on the memory aid as "Nausea"
Nausea - post dose 2 (Gastrointestinal disorders) | 7 (7) | 4/113 (4) — Solicited on the memory aid as "Nausea"
Injection site erythema, placebo arm - post dose 1 (General disorders) | 35 (35) | 55 (55) — Solicited on the memory aid as "Erythema (redness)" and measured in millimeters.
Injection site erythema, placebo arm - post dose 2 (General disorders) | 46 (46) | 60/113 (60) — Solicited on the memory aid as "Erythema (redness)" and measured in millimeters.
Injection site induration, placebo arm - (size) - post dose 1 (General disorders) | 16 (16) | 112 (112) — Solicited on the memory aid as "Induration (swelling)" and measured in millimeters.
Injection site induration, placebo arm - (size) - post dose 2 (General disorders) | 37 (37) | 111/113 (111) — Solicited on the memory aid as "Induration (swelling)" and measured in millimeters.
Injection site induration, placebo arm - (functional grading) - post dose 1 (General disorders) | 15 (15) | 113 (113) — Solicited on the memory aid as "Induration (swelling)" with grading based on impact on daily activities.
Injection site induration, placebo arm - (functional grading) - post dose 2 (General disorders) | 37 (37) | 110/113 (110) — Solicited on the memory aid as "Induration (swelling)" with grading based on impact on daily activities.
Injection site discolouration, placebo arm - post dose 1 (General disorders) | 1 (1) | 7 (7) — Solicited on the memory aid as "Pigmentation (discoloration)" and measured in millimeters.
Injection site discolouration, placebo arm - post dose 2 (General disorders) | 55 (55) | 3/113 (3) — Solicited on the memory aid as "Pigmentation (discoloration)" and measured in millimeters.
Injection site pain, placebo arm - post dose 1 (General disorders) | 14 (14) | 7 (7) — Solicited on the memory aid as "Pain at injection site at rest"
Injection site pain, placebo arm - post dose 2 (General disorders) | 16 (16) | 12/113 (12) — Solicited on the memory aid as "Pain at injection site at rest"
Tenderness, placebo arm - post dose 1 (General disorders) | 30 (30) | 16 (16) — Solicited on the memory aid as "Tenderness at injection site with movement/touch"
Tenderness, placebo arm - post dose 2 (General disorders) | 28 (28) | 21/113 (21) — Solicited on the memory aid as "Tenderness at injection site with movement/touch"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less